CLINICAL TRIAL: NCT06078163
Title: Combined Rehabilitation With ALA, ALC, Resveratrol and Vitamin D in Discogenic Sciatica in Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MFR0042023
Record Dates: First submitted 2023-09-28; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Sciatic Radiculopathy
MeSH Terms: interventions — Dietary Supplements; Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Treatment Group was composed of patients who will undergo daily pharmacological therapy with Alpha Lipoic Acid 600 mg, L-acetylcarnitine 1000 mg, Resvelatrol 50 mg, Vit D3 800UI for 30 consecutive days in combination with a rehabilitation protocol lasting 20 sessions
  Interventions: Other: supplementation; Other: rehabilitation
- Control Group (Placebo Comparator): Control Group was composed of patients who will only undergo a rehabilitation protocol lasting 20 sessions.
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: supplementation — daily pharmacological therapy with Alpha Lipoic Acid 600 mg, L-acetylcarnitine 1000 mg, Resvelatrol 50 mg, vit D3 800UI for 30 consecutive days in combination with a rehabilitation protocol lasting 20 sessions
  Arms: Treatment Group
Other: rehabilitation — rehabilitation protocol lasting 20 sessions.

SUMMARY:
The objective of this Interventional case-control clinical study is to evaluate the effectiveness of physiotherapy combined with the administration of Alpha Lipoic Acid, L-acetylcarnitine, Resvelatrol, Vit D3 in the treatment of sciatica due to herniated disc in young patients.

The main questions we intend to answer are:

* Is this combined treatment more effective in reducing pain?
* Is the combined treatment useful for improving postural alterations, reducing the intake of painkillers and the number of days of absence from work and improving the quality of life?

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years
* pain with NRS scale score between 5 and 7 points
* symptoms attributable to lumbosciatica which occurred no more than 4 weeks ago
* pharmacological wash out of NSAIDs and corticosteroids for at least a week
* presence of L4-L5, L5-S1 disc herniation diagnosed with lumbar MRI performed within 3 months
* absence of ongoing infectious episodes;
* written consent for participation in the study.

Exclusion Criteria:

* Altered states of consciousness;
* Sciatica not of disc origin
* Neurological disorders
* Presence of scoliosis >20° of Cobb
* Previous spinal surgery
* Pregnancy and/or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
extent of pain. | at the time of recruitment (T0); after 30 days from the start of treatment (T1); and after 60 days from the end of treatment (T2)
  Numeric Rating Scale (0-10)

SECONDARY OUTCOMES:
degree of disability of low back pain | at the time of recruitment (T0); after 30 days from the start of treatment (T1); and after 60 days from the end of treatment (T2)
  Oswestry Disability Questionnaire (ODQ) (0-50)
quality of life in relation to low back pain | at the time of recruitment (T0); after 30 days from the start of treatment (T1); and after 60 days from the end of treatment (T2)
  36-item Short Form Health Survey (SF-36) (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Functional Recovery and Rehabilitation Unit of the A.O.U.P. Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No